CLINICAL TRIAL: NCT04225962
Title: Intimacy of Women With Cystic Fibrosis
Acronym: IFAM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0422; 2019-A01988-49 (Other: ID-RCB)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Mucoviscidosis
Keywords: Cystic fibrosis; Women; Private life; Sexual disorders; Quality of sex life
MeSH Terms: conditions — Cystic Fibrosis; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with cystic fibrosis: Women with cystic fibrosis
  Interventions: Other: Intimate quality of life questionnaire

INTERVENTIONS:
Other: Intimate quality of life questionnaire — Preparation of an intimate quality of life questionnaire

SUMMARY:
The intimate life of patients with cystic fibrosis has not been the subject of specific research, it is even left behind in favor of respiratory, digestive or endocrinological dysfunctions endangering these patients. After 16 years of practice, it is significant that this subject is problematic, painful but difficult to tackle; No doubt just as much on the side of caregivers: this question has never found its way into team exchanges, it seems to be evaded doubtless difficult or too intimate to welcome. These disorders arise from the effects of the disease on the health of the mucous epithelial tissues also located in the genital area. These difficulties are more closely approached by the difficulties of procreation; PMA allows them to get around them, nevertheless making it possible to be a parent, with the residual frustration of a satisfactory sex life: a deaf "addition", adding to many care constraints.

It is therefore in terms of sexual health and quality of sexual life that it is desirable to shed light on this aspect of cystic fibrosis in women.

Bibliographic research confirms this approach: this subject is not explored, the rare publications concern the vulnerability of the cervix or the difficulty on both sides of tackling this subject.

ELIGIBILITY:
Inclusion Criteria:

* Major women with cystic fibrosis
* Tracked in the various CRCMs in France,
* Having or having had sexual intercourse,
* Having previously been informed of the aims and confidentiality of this research and not having opposed their participation.

Exclusion Criteria:

* Major women with cystic fibrosis whose state of health (acute episode of their disease or worsening phase) does not lend itself to such a collection
* Adult women with cystic fibrosis who are unable to receive the information and make a non-objection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Assessment of specific intimate disorders of patients with cystic fibrosis | 12 months
  Passing a questionnaire to assess patients' intimate quality of life.
  The responses to binary qualitative variables will be described by proportions. The responses to the 5-modality ordinal qualitative variables will be described by the median and the range (minimum and maximum). Continuous quantitative variables will be described by the mean and its standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise SIMONNET-BISSON, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud - CRCM adultes, médecine interne, Pierre-Bénite, France